CLINICAL TRIAL: NCT03874611
Title: Electrophysiology of Brain Activity During Electrode Implantation in Patients Treated With Deep Brain Stimulation
Acronym: LFP-DBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC11.242
Record Dates: First submitted 2018-04-30; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease; Obsessive-Compulsive Disorder; Epilepsy; Depression
MeSH Terms: conditions — Parkinson Disease; Obsessive-Compulsive Disorder; Epilepsy; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- electrophysiological data from DBS (Experimental)
  Interventions: Other: electrophysiological data from DBS

INTERVENTIONS:
Other: electrophysiological data from DBS — For each selected patient, the evaluation of cognitive or sensory-motor functions by electrophysiology will be conducted in the operating room, preoperatively the week before implantation and post-operatively within five days between the implantation of deep electrodes and the setting of the stimulator.

SUMMARY:
Primary objective

Demonstrate functional markers derived from electrophysiological signals recorded during cognitive tests. These markers should make it possible to optimize the targeting procedures of electrode implantation sites for a better effectiveness of deep brain stimulation therapy.

Research hypotheses

The mechanisms of action of the deep brain stimulation (DBS) involve the modulation of the activity, locally and on a large scale, of functional cortical-subcortical networks showing pathological behavior beforehand. The electrophysiological measurements in response to different tasks make it possible to highlight precise dysfunctions of these neural networks, in relation with the behavioral and / or motor disorders associated with the pathologies treated by DBS.

Consequently, we hypothesize that the exploitation of electrophysiological responses during cognitive or sensorimotor tasks performed during the implantation procedure of stimulation electrodes in patients treated with DBS will allow :

* To collect fundamental data to understanding the physiological functioning of basal ganglia in humans ;
* To collect functional markers from the operating room in relation to the symptoms targeted by the DBS that will help in the choice of implantation site of the stimulation electrode ;
* Define long-term predictive markers of DBS effects by comparing electrophysiological effects measured post-operatively and clinical scores under DBS.

ELIGIBILITY:
Inclusion Criteria:

* Pathology requiring brain stimulation therapy (criteria of severity, therapeutic resistance and severity of disability): motor disorders (eg Parkinson's disease, dystonia) or psychiatric disorders (eg OCD, depression).
* These pathologies therefore include motor disorders (eg Parkinson's disease, dystonia) or psychiatric disorders that can be treated with brain stimulation therapy. Note that these are independent of motor disorders. The inclusion criteria obviously depend on the pathology.

As an example for a motor pathology treated by stimulation, in Parkinson's disease the following inclusion criteria are used :

* patients aged 18 to 75 and affiliated to a social security scheme
* Idiopathic Parkinson's disease that meets the United Kingdom Parkinson's Disease Brain Bank (UKPDSBB) criteria or suffering from recessive autosomal juvenile parkinsonism
* duration of evolution of the disease> 5 years
* stage of severe motor complications of levodopa despite optimal treatment.

For dystonic patients, the following inclusion criteria are used :

* Disabling dystonia (severe focal, segmental or generalized).
* Patient ≥ 18 years of age and under age 65
* Duration of evolution of dystonia greater than one year.

For patients with obsessive-compulsive disorder (OCD), the following inclusion criteria are used :

* OCD which has been diagnosed for at least 5 years according to the DSM-IV criteria as OCD with "good insight", confirmed using the Diagnostic Interview Genetic Study (DIGS) - OCD section ; score below the delusional idea threshold at the BABS (Brown Assessment of Beliefs Scale) insight scale (Eisen, Phillips et al., 1998)
* OCD of severe intensity (total YBOCS > 25, or subscale Obsessions or Compulsions > 15, EGF < 40, CGI > 4) with prognosis considered to be bad in the absence of intervention
* Non-responder OCD (an improvement of less than 25% on the Y-BOCS scale) to at least three IRS-type antidepressants, including clomipramine, used sequentially at the maximum tolerated dose for at least 12 weeks. Used alone and in combination for at least 1 month with risperidone or pimozide and any of the following products : lithium salts or clonazepam or buspirone or pindolol (Greist and Jefferson 1998) (McDougle, Epperson et al 2000) (Dannon , Sasson et al., 2000)
* OCD having benefited from Behavioral and Cognitive Therapy for at least 1 year (application of classical programs, including exposure techniques with prevention of ritualized response, with at least two sessions per month).
* Patient between 18 and 60 years of age who has given his signature and informed consent after receiving written information on the proposed procedure
* Sick with social security

For patients with depressive illness, the following inclusion criteria were used :

* male or female between the ages of 30 and 65
* with a diagnosis of unipolar major depression (MINI) resistant to conventional treatments
* Hamilton and Montgomery Depression Scale (HAMD) score> 20
* Duration of the current depressive episode of more than 12 months, the patient being included in a care system has established the chronic and recurrent state of this depression,
* Ineffective treatment of the current episode with at least 4 therapeutic attempts including antidepressant drug monotherapy treatments (MAOIs, tricyclic antidepressants, selective serotonin reuptake inhibitors, mixed serotonin reuptake inhibitors, and norepinephrine), the potentiations of antidepressant treatments (by lithium salts, thyroid hormones or neuroleptics), the psychotherapies structured according to validated techniques, the ECT carried out under conditions in conformity with the recommendations (ANAES, 1998) (at least 6 sessions in technical bilateral with control of duration of seizure)

  * Women of childbearing age should follow a contraceptive method that is considered sufficiently effective by the investigator. In this case a pregnancy test will be performed on inclusion
  * outpatient or inpatient
  * fluent in the French language and able to understand the procedures of the study and in particular complete the self-questionnaires used
  * Patient likely to give informed consent
  * Patient affiliated with Social Security
  * Patient's written agreement to participate in the study
  * Intellectual abilities compatible with cognitive or motor tasks

Exclusion Criteria:

* Persons referred to in Articles L1121-5 to L1121-8 of the CSP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2011-04-13 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of functional markers derived from electrophysiological signals recorded during cognitive tests. | 5 days
  The latency of task-related electrophysiological responses derived from deep brain electrodes, as assessed by time-frequency and evoked-responses analyses.
Number of functional markers derived from electrophysiological signals recorded during cognitive tests. | 5 days
  The amplitude of task-related electrophysiological responses derived from deep brain electrodes, as assessed by time-frequency and evoked-responses analyses.

SECONDARY OUTCOMES:
cognitive and sensorimotor tasks | 5 days
  percentage of electrode contacts within a given brain area that will display task-evoked neural responses (as assessed by time-frequency analyses) for a given task.
functional atlas of basal ganglia | 5 days
  statistical effects of each task as assessed by t-tests performed across patient's task-related electrophysiological responses (as assessed by time-frequency analyses).
number of electrophysiological responses | 5 days
  time and frequency analyses

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No